CLINICAL TRIAL: NCT00928668
Title: Randomised, Double-Blind, Placebo-Controlled, 5-Way Cross-Over Study to Assess the Efficacy (Bronchoprotection) and Safety of a Single Dose of Orally Inhaled BI 1744 CL (2, 5, 10 and 20ug) in Patients With Intermittent Asthma
Brief Title: Efficacy (Bronchoprotection) and Safety of Orally Inhaled BI 1744 CL in Patients With Intermittent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.4
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — olodaterol

ARMS (5):
- Olodaterol (BI1744) Low (Experimental): Single dosing of low dose Olodaterol inhaled orally from Respimat Device
  Interventions: Drug: Olodaterol (BI1744CL)
- Olodaterol (BI1744) Medium Low (Experimental): Single dosing of medium low dose Olodaterol inhaled orally from Respimat Device
  Interventions: Drug: Olodaterol (BI1744CL)
- Olodaterol (BI1744) Medium High (Experimental): Single dosing of medium high dose Olodaterol inhaled orally from Respimat Device
  Interventions: Drug: Olodaterol (BI1744CL)
- Olodaterol (BI 1744) High (Experimental): Single dosing of high dose Olodaterol inhaled orally from Respimat Device
  Interventions: Drug: Olodaterol (BI1744CL)
- Placebo (Placebo Comparator): Single dosing of Olodaterol placebo inhaled orally from Respimat Device
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo device for comparison
  Arms: Placebo
Drug: Olodaterol (BI1744CL) — Olodaterol comparison of low, medium low, medium high and high doses
  Arms: Olodaterol (BI1744) Medium High
Drug: Olodaterol (BI1744CL) — Olodaterol comparison of low, medium low, medium high and high doses
  Arms: Olodaterol (BI1744) Low
Drug: Olodaterol (BI1744CL) — Olodaterol comparison of low, medium low, medium high and high doses
  Arms: Olodaterol (BI1744) Medium Low
Drug: Olodaterol (BI1744CL) — Olodaterol comparison of low, medium low, medium high and high doses
  Arms: Olodaterol (BI 1744) High

SUMMARY:
The primary objective of this study is to assess the efficacy (bronchoprotection) and safety of single doses of BI 1744 CL inhalation solution (2, 5, 10 and 20 mcg) delivered via the Respimat® inhaler, in patients with intermittent asthma.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of intermittent asthma according to Global Initiative for Asthma criteria
2. Non-smokers or ex-smokers who have not smoked for at least 1 year and have a smoking history of less than 5 pack-years
3. Forced Expiratory Volume in 1second greater than or equal to 80% predicted normal (Visit 1).
4. Bronchial hyperresponsiveness to inhaled methacholine with a provocative concentration of a methacholine causing a 20% fall in Forced Expiratory Volume in one second less than or equal to 8 mg/mL (Visit 1).
5. Be able to perform technically acceptable pulmonary function tests
6. Be able to inhale medication in a competent manner from the Respimat® inhaler
7. Must sign and date an informed consent consistent with International Conference on Harmonisation-Good Clinical Practice guidelines prior to participation in the trial, which includes medication washout and restrictions.

Exclusion criteria

1. Patients with a significant disease other than asthma
2. Patients with seasonal asthma or allergies whose participation in the trial will occur during the season for which they are allergic.
3. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis; all patients with a serum glutamic oxaloacetic transaminase > 80 IU/L, serum glutamic pyruvic transaminase > 80 IU/L, bilirubin >2.0 mg/dL or creatinine > 2.0 mg/dL will be excluded regardless of clinical condition
4. Patients with any of the following conditions: a diagnosis of hyperthyrosis or paroxysmal tachycardia (>100 beats per minute), a marked baseline prolongation of QT/QTc interval, a history of additional risk factors for Torsade de Pointes, a history of myocardial infarction, a diagnosis of clinically relevant cardiac arrhythmia, a history of cor pulmonale, known active tuberculosis, a malignancy for which the patient has undergone resection, radiation therapy or chemotherapy within the last five years (patients with treated basal cell carcinoma are allowed), a history of life-threatening pulmonary obstruction, a history of cystic fibrosis, clinically evident bronchiectasis, or a history of significant alcohol or drug abuse.
5. Patients who have undergone thoracotomy with pulmonary resection
6. Patients who are being treated with any of the following concomitant medications: medications that prolong the QT/QTc interval, oral beta-adrenergics, beta-blockers or monoamine oxidase inhibitors or tricyclic antidepressants.
7. Patients who have been treated with any respiratory medications (excluding short-acting beta-agonists) for control of their asthma symptoms within 3 months of the Screening Visit (Visit 1).
8. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit (Visit 1).
9. Pregnant or nursing women, or women of childbearing potential not using a highly effective method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-01; Primary Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Canada (4):
  - 1222.4.103 UBC - Respiratory Medicine, Vancouver, British Columbia
  - 1222.4.104 Department of Medicine, Health Sciences Centre, Hamilton, Ontario
  - 1222.4.101 2725 Chemin Ste Foy, Sainte-Foy, Quebec
  - 1222.4.102, Saskatoon, Saskatchewan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, placebo-controlled, 5-way crossover trial. The duration of each treatment period was 1 day with a 14 day washout period between treatments.
Pre-assignment Details: One patient was randomized, but the trial was put on hold so that the patient had to be discontinued and re-randomized. This causes a discrepancy between the 32 patients enrolled and the 31 patients reported for the participant flow.
Groups:
- Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg: Patients were administered Olodaterol 5 mcg qd in the first period, Olodaterol 2 mcg qd in the second period, Olodaterol 10 mcg qd in the third period, matching Placebo in the fourth period and Olodaterol 20 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 10mcg / Olo 20mcg / Olo 2mcg / Olo 5mcg / Placebo: Patients were administered Olodaterol 10 mcg qd in the first period, Olodaterol 20 mcg qd in the second period, Olodaterol 2 mcg qd in the third period, Olodaterol 5 mcg qd in the fourth period and matching Placebo in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 2mcg / Placebo / Olo 20mcg / Olo 10mcg / Olo 5mcg: Patients were administered Olodaterol 2 mcg qd in the first period, matching Placebo in the second period, Olodaterol 20 mcg qd in the third period, Olodaterol 10 mcg qd in the fourth period and Olodaterol 5 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg / Olo 10mcg: Patients were administered Olodaterol 20 mcg qd in the first period, Olodaterol 5 mcg qd in the second period, matching Placebo in the third period, Olodaterol 2 mcg qd in the fourth period and Olodaterol 10 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
- Placebo / Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg: Patients were administered matching Placebo in the first period, Olodaterol 10 mcg qd in the second period, Olodaterol 5 mcg qd in the third period, Olodaterol 20 mcg qd in the fourth period and Olodaterol 2 mcg qd in the fifth period. Olodaterol was administered via the Respimat inhaler.
Period: Overall Study
Arm/Group | Olo 5mcg / Olo 2mcg / Olo 10mcg / Placebo / Olo 20mcg | Olo 10mcg / Olo 20mcg / Olo 2mcg / Olo 5mcg / Placebo | Olo 2mcg / Placebo / Olo 20mcg / Olo 10mcg / Olo 5mcg | Olo 20mcg / Olo 5mcg / Placebo / Olo 2mcg / Olo 10mcg | Placebo / Olo 10mcg / Olo 5mcg / Olo 20mcg / Olo 2mcg
Started | 7 | 7 | 7 | 4 | 6
Completed | 6 | 6 | 6 | 3 | 5
Not Completed | 1 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Other reasons not listed above | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Total: Total number of patients treated in the study. This was a randomised, double-blind, placebo-controlled, 5-way crossover trial. 31 patients were assigned randomly to one of 5 treatment sequences in which they received each of 5 treatments. The duration of each treatment period was 1 day with a 14 day washout period between treatments.
Arm/Group | Study Total
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean of Provocative Concentration of Methacholine Required to Produce a 20% Decrease in FEV1 (PC20FEV1) at 24 Hours
Description: Provocative concentration of methacholine required to produce a 20% decrease in FEV1 (PC20FEV1) at 24 hours
Time Frame: 24 hours post dose
Population: Full analysis set (FAS). FAS is defined as all patients that were randomised, received treatment and had baseline data and post-dose data for at least two periods for the same endpoint.
Measure: Least Squares Mean (Standard Error); unit: Log base 2 (mg/ml)
Groups:
- Placebo: Matching Placebo delivered by the Respimat Inhaler.
- Olodaterol (Olo) 2 mcg qd: Olodaterol 2 mcg qd delivered by the Respimat Inhaler.
- Olodaterol (Olo) 5 mcg qd: Olodaterol 5 mcg qd delivered by the Respimat Inhaler.
- Olodaterol (Olo) 10 mcg qd: Olodaterol 10 mcg qd delivered by the Respimat Inhaler.
- Olodaterol (Olo) 20 mcg qd: Olodaterol 20 mcg qd delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olodaterol (Olo) 2 mcg qd | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Olodaterol (Olo) 20 mcg qd
Number analyzed (Participants) | 29 | 28 | 27 | 30 | 29
Log base 2 (mg/ml) | 0.793 (0.182) | 1.950 (0.186) | 2.504 (0.190) | 3.236 (0.179) | 3.777 (0.183)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Adjusted using an analysis of variance with terms for centre, patients within centre, treatment and period (all as fixed effects); Mean Difference (Final Values) = 1.157, 95% CI 2-sided [0.657 to 1.657], Standard Error of Mean 0.252 — Olo 2 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.711, 95% CI 2-sided [1.205 to 2.217], Standard Error of Mean 0.255 — Olo 5 mcg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.443, 95% CI 2-sided [1.952 to 2.935], Standard Error of Mean 0.248 — Olo 10 mcg minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olodaterol (Olo) 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.984, 95% CI 2-sided [2.486 to 3.483], Standard Error of Mean 0.251 — Form 20 mcg minus Placebo

2. Secondary Outcome: Adjusted Mean of Provocative Concentration of Methacholine Required to Produce a 20% Decrease in FEV1 (PC20FEV1) at 30 Minutes
Description: Provocative concentration of methacholine required to produce a 20% decrease in FEV1 (PC20FEV1) at 30 minutes
Time Frame: 30 minutes post dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Log base 2 (mg/ml)
Arm/Group | Placebo | Olodaterol (Olo) 2 mcg qd | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Olodaterol (Olo) 20 mcg qd
Number analyzed (Participants) | 29 | 28 | 27 | 30 | 29
Log base 2 (mg/ml) | 0.393 (0.180) | 2.532 (0.184) | 3.029 (0.187) | 3.953 (0.177) | 4.617 (0.181)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.139, 95% CI 2-sided [1.645 to 2.633], Standard Error of Mean 0.249 — Olo 2 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.636, 95% CI 2-sided [2.135 to 3.136], Standard Error of Mean 0.252 — Olo 5 mcg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.560, 95% CI 2-sided [3.074 to 4.046], Standard Error of Mean 0.245 — Olo 10 mcg minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olodaterol (Olo) 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.224, 95% CI 2-sided [3.731 to 4.717], Standard Error of Mean 0.249 — Form 20 mcg minus Placebo

3. Secondary Outcome: Adjusted Mean of Provocative Concentration of Methacholine Required to Produce a 20% Decrease in FEV1 (PC20FEV1) at 4 Hours
Description: Provocative concentration of methacholine required to produce a 20% decrease in FEV1 (PC20FEV1) at 4 hours
Time Frame: 4 hours post dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Log base 2 (mg/ml)
Arm/Group | Placebo | Olodaterol (Olo) 2 mcg qd | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Olodaterol (Olo) 20 mcg qd
Number analyzed (Participants) | 29 | 28 | 27 | 30 | 29
Log base 2 (mg/ml) | 0.577 (0.214) | 2.602 (0.219) | 2.957 (0.223) | 4.126 (0.211) | 4.786 (0.215)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.025, 95% CI 2-sided [1.437 to 2.613], Standard Error of Mean 0.296 — Olo 2 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.380, 95% CI 2-sided [1.785 to 2.975], Standard Error of Mean 0.300 — Olo 5 mcg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.549, 95% CI 2-sided [2.971 to 4.127], Standard Error of Mean 0.292 — Olo 10 mcg minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olodaterol (Olo) 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.208, 95% CI 2-sided [3.622 to 4.794], Standard Error of Mean 0.296 — Form 20 mcg minus Placebo

4. Secondary Outcome: Adjusted Mean of Provocative Concentration of Methacholine Required to Produce a 20% Decrease in FEV1 (PC20FEV1) at 8 Hours
Description: Provocative concentration of methacholine required to produce a 20% decrease in FEV1 (PC20FEV1) at 8 hours
Time Frame: 8 hours post dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Log base 2 (mg/ml)
Arm/Group | Placebo | Olodaterol (Olo) 2 mcg qd | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Olodaterol (Olo) 20 mcg qd
Number analyzed (Participants) | 29 | 28 | 27 | 30 | 29
Log base 2 (mg/ml) | 0.576 (0.213) | 2.484 (0.218) | 3.050 (0.222) | 3.903 (0.210) | 4.796 (0.214)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.907, 95% CI 2-sided [1.322 to 2.492], Standard Error of Mean 0.295 — Olo 2 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.474, 95% CI 2-sided [1.822 to 3.066], Standard Error of Mean 0.299 — Olo 5 mcg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.327, 95% CI 2-sided [2.752 to 3.902], Standard Error of Mean 0.290 — Olo 10 mcg minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olodaterol (Olo) 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.220, 95% CI 2-sided [3.637 to 4.803], Standard Error of Mean 0.294 — Form 20 mcg minus Placebo

5. Secondary Outcome: Adjusted Mean of Provocative Concentration of Methacholine Required to Produce a 20% Decrease in FEV1 (PC20FEV1) at 32 Hours
Description: Provocative concentration of methacholine required to produce a 20% decrease in FEV1 (PC20FEV1) at 32 hours
Time Frame: 32 hours post dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Log base 2 (mg/ml)
Arm/Group | Placebo | Olodaterol (Olo) 2 mcg qd | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Olodaterol (Olo) 20 mcg qd
Number analyzed (Participants) | 28 | 28 | 27 | 30 | 29
Log base 2 (mg/ml) | 0.960 (0.200) | 2.189 (0.200) | 2.785 (0.203) | 3.074 (0.192) | 3.605 (0.197)
Statistical Analysis 1: Comparison: Placebo vs Olodaterol (Olo) 2 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.229, 95% CI 2-sided [0.692 to 1.766], Standard Error of Mean 0.271 — Olo 2 mcg minus Placebo
Statistical Analysis 2: Comparison: Placebo vs Olodaterol (Olo) 5 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.825, 95% CI 2-sided [1.281 to 2.369], Standard Error of Mean 0.274 — Olo 5 mcg minus Placebo
Statistical Analysis 3: Comparison: Placebo vs Olodaterol (Olo) 10 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.114, 95% CI 2-sided [1.578 to 2.650], Standard Error of Mean 0.270 — Olo 10 mcg minus Placebo
Statistical Analysis 4: Comparison: Placebo vs Olodaterol (Olo) 20 mcg qd; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.645, 95% CI 2-sided [2.110 to 3.181], Standard Error of Mean 0.270 — Form 20 mcg minus Placebo

6. Secondary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG
Description: Clinical relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinalysis and ECG. New abnormal findings or worsenings of baseline conditions were reported as Adverse Events (cardiac disorders and investigations).
Time Frame: 5 days
Population: The safety set included all patients who received any study medication.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Matching Placebo delivered by the Respimat resp. Aerolizer Inhaler.
- Olo 2 mcg: Olodaterol 2 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 5 mcg: Olodaterol 5 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 10 mcg: Olodaterol 10 mcg qd (morning) delivered by the Respimat Inhaler.
- Olo 20 mcg: Olodaterol 20 mcg qd delivered by the Respimat Inhaler.
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Number analyzed (Participants) | 29 | 28 | 28 | 30 | 29
percentage of participants
  Cardiac disorders | 0 | 0 | 0 | 0 | 0
  Investigations | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Laboratory Testing: Average Change From Baseline of Potassium and Calcium
Description: Laboratory testing: Average change from baseline of potassium and calcium measured on test-days
Time Frame: Baseline to Visit 6
Population: All patients in the Safety set who have a baseline value and post dose values for each planned time.
Measure: Geometric Mean (Inter-Quartile Range); unit: mmol/L
Arm/Group | Placebo | Olodaterol (Olo) 2 mcg qd | Olodaterol (Olo) 5 mcg qd | Olodaterol (Olo) 10 mcg qd | Olodaterol (Olo) 20 mcg qd
Number analyzed (Participants) | 29 | 26 | 26 | 29 | 28
mmol/L
  Potassium | 1.01 (NA) [0.98 to 1.05] | 1.04 (NA) [1.00 to 1.06] | 1.02 (NA) [1.00 to 1.05] | 1.00 (NA) [0.98 to 1.03] | 0.98 (NA) [0.95 to 1.02]
  Calcium | 1.00 (NA) [0.98 to 1.03] | 1.01 (NA) [0.99 to 1.02] | 1.00 (NA) [0.98 to 1.03] | 1.00 (NA) [0.99 to 1.02] | 1.01 (NA) [0.99 to 1.03]

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Single dose including washout phase
Arm/Group | Placebo | Olo 2 mcg | Olo 5 mcg | Olo 10 mcg | Olo 20 mcg
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28 | 0/28 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 4/29 | 1/28 | 1/28 | 1/30 | 4/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Olo 2 mcg (N=28) | Olo 5 mcg (N=28) | Olo 10 mcg (N=30) | Olo 20 mcg (N=29)
Headache (Nervous system disorders) | 3 | 0 | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication